CLINICAL TRIAL: NCT05268445
Title: Comparison of Two Validated Endovascular Strategies for Refractory Vasospastic Stenosis After Non-traumatic Intracranial Haemorrhage Leading to Severe Brain Hypoperfusion: Chemical Versus Chemical and Mechanical Angioplasty
Brief Title: Chemical and Mechanical Angioplasty for Vasospasm (SAVEBRAIN)
Acronym: SAVEBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRB2021297
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Vasospasm, Intracranial; Stenosis; Ruptured Cerebral Aneurysm; Arteriovenous Malformations, Cerebral; Arteriovenous Fistula
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Constriction, Pathologic; Intracranial Arteriovenous Malformations; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: Randomization between chemical angioplasty and chemical plus mechanical angioplasty using an adjustable remodeling mesh or a balloon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemical angioplasty (Active Comparator): Chemical angioplasty using intra-arterial Nimodipin
  Interventions: Procedure: Chemical and Mechanical Angioplasty for Refractory Intracranial Arterial Vasospastic Stenosis
- Chemical and Mechanical angioplasty (Active Comparator): Balloon angioplasty for refractory intracranial arterial vasospastic stenosis with a CE Marked device (Neurospeed balloon) or Adjustable remodeling mesh angioplasty for refractory intracranial arterial vasospastic stenosis with a CE Marked device (Comaneci) in association with intra-arterial Nimodipin
  Interventions: Procedure: Chemical and Mechanical Angioplasty for Refractory Intracranial Arterial Vasospastic Stenosis

INTERVENTIONS:
Procedure: Chemical and Mechanical Angioplasty for Refractory Intracranial Arterial Vasospastic Stenosis — Angioplasty for Refractory Intracranial Arterial Vasospastic Stenosis

SUMMARY:
This is a monocentric randomized prospective trial comparing 2 different endovascular strategies of intracranial arterial angioplasty in case of refractory intracranial arterial vasospastic stenosis :

* chemical angioplasty
* chemical and mechanical angioplasty

DETAILED DESCRIPTION:
Compare in a randomized prospective trial 2 approved treatments of refractory intracranial arterial vasospastic stenosis, chemical angioplasty versus chemical and mechanical angioplasty, using devices already used in clinical practice and CE marked: chemical angioplasty using Nimotop versus chemical and mechanical angioplasty with balloon or adjustable remodeling mesh on brain perfusion evaluated by brain computed tomography (CT) Perfusion

Nowadays, the choice between chemical or chemical and mechanical angioplasty depends on the neurointerventionist for each procedure, no difference in efficiency or safety has been proved and no solid scientific data helps the physician in choosing the correct treatment for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Non-traumatic intracranial hemorrhage (ruptured aneurysm, AVM, or per-procedural complication etc)
3. Ruptured aneurysm, AVM, intracranial arterial perforation or any bleeding lesion secured with surgical clipping or endovascular intervention.
4. No contra-indication to both CTP and MRI imaging
5. Subject or legal representative is able and willing to give informed consent.
6. Refractory of intracranial arterial vasospastic stenosis requiring an endovascular angioplasty with a severe stenosis defined on CTA or DSA; and/or a significant hypoperfusion defined according to the mismatch profile in stroke or a MTT>6 seconds. The volume of critically hypoperfused tissue will be based on a time to maximum of the tissue residue function (Tmax) threshold of >6 sec using the Rapid (or equivalent) software.

Exclusion Criteria:

1. Angioplasty by one of the two methods considered as impossible or too risky by the neurointerventionist
2. Inability to obtain consent from patient or patients relatives
3. Pregnant women
4. Less than 18 years of age
5. Need to use any other device
6. Vertebro-basilar arteries will not be randomized because of the difficulty to assess the perfusion volume in this territory, but will be treated if necessary according to our local protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in brain hypoperfusion | Change between day 0 and day 1 after the endovascular procedure and randomization
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion Time to drain (seconds) on CT and/or MR perfusion

SECONDARY OUTCOMES:
Change in vessel size | Change between day 0 and day 1 after the endovascular procedure and randomization
  Change in the vessel size measured on digital subtraction angiography (DSA) and computed tomography angiogram (CTA) in millimeters
Time to next endovascular intervention for vasospastic stenosis | Number of days after the endovascular procedure until the next procedure in days, up to 4 weeks
  Delay between two procedures for the same indication
modified Rankin Scale at 3 months | 3 months after Intracranial Hemorrhage
  clinical evolutionclinical evolution (mRS between 0 and 6, a higher score means a worse outcome)
Change in Transcranial Doppler | Change between day 0 and day 1 after the endovascular procedure and randomization
  Change in intracranial vasospasm assessed by the targeted vessel velocity in meters per second
change in Brain Hypoperfusion 2 | Change between day 0 and day 1 after the endovascular procedure and randomization
  Reduction in brain hypoperfusion assessed by the volumes on different perfusion parameters time to peak (in seconds) on CT and/or MR perfusion
change in Glasgow coma scale | Change between day 0 and day 1 after the endovascular procedure and randomization
  Glasgow coma scale (GCS between 3 and 15, a higher score means a better outcome)
change in National Institutes of Health Stroke Scale score | Change between day 0 and day 1 after the endovascular procedure and randomization
  National Institutes of Health Stroke Scale (NIHSS between 0 and 42, a higher score means a worse outcome)
Change in the monitoring of tissue oxygen pressure (PtiO2) | Change between day 0 and day 1 after the endovascular procedure and randomization
  Monitoring of tissue oxygen pressure (PtiO2)
Number of new ischemic lesions | Change between day 0, 5, 9, 21 after Intracranial Hemorrhage
  Number of new ischemic lesions on non-contrast computed tomography (CT) scan
Change in brain hypoperfusion 3 | Change between day 0 and day 1 after the endovascular procedure and randomization
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion parameters TMax maps in seconds on CT and/or MR perfusion
Change in brain hypoperfusion 4 | Change between day 0 and day 1 after the endovascular procedure and randomization
  Brain hypoperfusion in arterial territories assessed by the delays on perfusion parameters Mean transit time on CT and/or MR perfusion in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Guenego, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD sharing